CLINICAL TRIAL: NCT00549822
Title: A Phase II Clinical Trial of Intermittent Letrozole Therapy in Postmenopausal Women With CA 15-3 Positive (Carcinoma Antigen 15-3), Hormone Receptor Positive, Metastatic Breast Cancer
Brief Title: Intermittent Letrozole Therapy in Postmenopausal Women With Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Novartis (Industry)
Responsible Party: Principal Investigator, Paul Goss, MD, PhD, Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-109
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: aromatase inhibitor; CA 15-3; Hormone receptor positive
MeSH Terms: conditions — Breast Neoplasms; Medullary cystic kidney disease 1 | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intermittent letrozole therapy (Experimental): Letrozole 2.5 mg administered by mouth daily during each 28 day treatment cycle. Treatment is intermittent with possible breaks between each 28 day treatment cycle based on CA 15-3 or CA 27.29 levels. Letrozole is administered until the participant has disease progression as determined by RECIST (Response Evaluation Criteria In Solid Tumors), experiences severe side effects, or decides to stop treatment.
  Interventions: Drug: Letrozole

INTERVENTIONS:
Drug: Letrozole — Treatment is intermittent with possible breaks between each 28 day treatment cycle if CA 15-3 or CA 27.29 level that has decreased by at least 50% of that individual patient's baseline or peak level on firstline letrozole or anastrozole therapy or has decreased into the normal reference range per institutional parameters. Letrozole or anastrozole therapy will be interrupted until CA 15-3 or CA 27.29 levels rise by at least 25% above trough CA 15-3 or CA 27.29 level. If the trough level is in the normal reference range then the CA 15-3 or CA 27.29 must rise into the normal reference range.
  Other Names: Femara

SUMMARY:
The purpose of this research study is to study the effects of using aromatase inhibitor (AI) therapy intermittently on participants with breast cancer. AIs are a class of drugs used to treat breast cancer in postmenopausal women. They work by decreasing the level of estrogen, which is believed to stimulate the growth of tumor tissue. Breast cancer that progresses despite therapy with an AI is thought to have become resistant to AI therapy. There is scientific evidence to suggest that resistant breast cancer cells learn to grow at the very low levels of estrogen present on AI therapy, and that increasing estrogen levels even slightly by stopping AI therapy may inhibit the breast cancer cells.

DETAILED DESCRIPTION:
* This study involves treating participants with intermittent AI therapy. The AI will be stopped at the time they enter the study. We plan on monitoring a marker in the participants blood called CA 15-3 (or CA 27.29) every 4 weeks to help us make a decision of when to re-start treatment with letrozole (femara). This marker is known to rise when disease is progressing and drop when the disease is responding to treatment. We will be stopping and re-starting therapy based on the changes of CA 15-3 in the participants blood.
* In addition to bloodwork, the following tests and procedures will be performed on a monthly basis: medical history; physical examination and performance status.
* Every 8 weeks the following will be performed: Tumor assessment by physical exam (if possible); Chest x-ray or CT scan or chest; CT scans of abdomen and pelvis; and bone scan.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18 years of age or older
* Postmenopausal
* Histologically or cytologically confirmed adenocarcinoma of the breast with locally advanced or metastatic disease this is not considered amenable to curative treatment with elevation of CA 15-3 documented at the time of diagnosis of metastatic disease and prior to initiation of letrozole or anastrozole therapy
* Current letrozole or anastrozole monotherapy with a documented CA 15-3 level that has decreased by at least 50% of the patients baseline
* Letrozole or anastrozole must be discontinued at the time of study enrollment
* Evidence of hormone sensitivity of primary or secondary tissue.
* Measurable or nonmeasurable (but evaluable-defined as nontarget lesions) disease according to modified RECIST
* Prior antiestrogen therapies including tamoxifen, steroidal AIs, nonsteroidal AIs, or fulvestrant in the adjuvant setting is allowed provided the patient is currently on letrozole or anastrozole monotherapy as first-line therapy for metastatic disease
* Life expectancy of greater than 3 months
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0,1, or 2
* Normal organ and marrow function as outlined in protocol

Exclusion Criteria:

* Premenopausal
* Trastuzumab or biologic therapy within 2 weeks
* Prior or planned radiation therapy to a site of evaluable disease in the event that the site is the only site of evaluable disease
* Concomitant anticancer treatments including trastuzumab, chemotherapy, or other biologic agents other than letrozole or anastrozole therapy
* Chronic bisphosphonates for hypercalcemia or prevention of bone metastases.
* Treatment with non-approved or investigational agent within 2 weeks before study entry
* Presence of life-threatening metastatic disease, defined as extensive hepatic involvement, or past or present brain or leptomeningeal involvement, or symptomatic pulmonary lymphangitic spread
* Patients who are highly symptomatic from their breast cancer, or who require urgent palliative chemotherapy, as decided by their treating physician
* Previous or current systemic malignancy within the past five years, except for contralateral breast carcinoma, in situ carcinoma of the cervix treated by cone biopsy, or adequately treated basal or squamous cell carcinoma of the skin.
* Any severe concomitant condition believed to render subject undesirable for participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2007-10 (Actual); Primary Completion 2010-05 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Goss, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postmenopausal patients with ER-positive (ER+) metastatic breast cancer (MBC) that were enrolled on an institutional review board (IRB) approved, phase II, multicenter clinical trial protocol (NCT00549822) evaluating intermittent AI (Aromatase Inhibitor) therapy. The study opened to accrual August 29, 2006 and closed to accrual on May 17, 2010.
Groups:
- Intermittent Letrozole Therapy: Letrozole 2.5mg: Intermittently
  Letrozole 2.5 mg administered by mouth each day during each 28 day treatment cycle. Treatment is intermittent with possible breaks between each 28 day treatment cycle. Letrozole is administered until the participant has disease progression as determined by RECIST (Response Evaluation Criteria In Solid Tumors), experiences severe side effects, or decides to stop treatment.
Period: Overall Study
Arm/Group | Intermittent Letrozole Therapy
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intermittent Letrozole Therapy
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Decline in Serum CA 15-3 (Carcinoma Antigen 15-3)
Description: The Number of patients that have have a response of a decrease in CA 15-3 or CA 27.29 levels by at least 50% of that individual patient's baseline or peak level after re-introducing Letrozole therapy following a break in therapy as described in the intervention.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Intermittent Letrozole Therapy
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Median Time to Disease Progression With Intermittent Letrozole.
Description: The median time to disease progression as determined by RECIST (Response Evaluation Criteria In Solid Tumors).
Time Frame: 3 years
Measure: Median (Full Range); unit: Months
Arm/Group | Intermittent Letrozole Therapy
Number analyzed (Participants) | 3
Months | 47 [28.5 to NA] — Third participant did not have progressive disease during study follow-up.

3. Secondary Outcome: Serum HER-2/Neu Levels and Serum/Plasma Angiogenic Mediators
Description: Measurements for the serum HER-2/neu (human epidermal growth factor receptor 2) levels and serum/plasma angiogenic mediators
Time Frame: 2 years
Population: Study terminated prematurely due to slow accrual. Outcome measure data not available for analysis.
Arm/Group | Intermittent Letrozole Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Duration of treatment and twelve weeks after stopping treatment.
Description: Adverse events are recorded when reported by subjects and systematically evaluated through laboratory tests, physicals, and physician interviews every four weeks for the duration of treatment. Patients are followed for 12 weeks after removal from study or until death, whichever occurs first.
Groups:
- Intermittent Letrozole Therapy: Letrozole 2.5mg: Intermittently
Arm/Group | Intermittent Letrozole Therapy
All-Cause Mortality (participants affected / at risk) | 2/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intermittent Letrozole Therapy (N=3)
Hemoglobin (Blood and lymphatic system disorders) | 2 (24)
Lymphopenia (Blood and lymphatic system disorders) | 1 (12)
Fatigue (General disorders) | 3 (54)
Weight loss (General disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Skin-other (Skin and subcutaneous tissue disorders) | 1 (2)
Hot flashes (Endocrine disorders) | 3 (54)
Constipation (Gastrointestinal disorders) | 3 (54)
Gastritis (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 3 (54)
Hemorrhage-other (Blood and lymphatic system disorders) | 1 (13)
Infection Gr0-2 neut, sinus (Infections and infestations) | 1 (1)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (5)
ALT, SGPT (Metabolism and nutrition disorders) | 1 (6)
AST, SGOT (Metabolism and nutrition disorders) | 1 (6)
Creatinine (Metabolism and nutrition disorders) | 1 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (14)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3)
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 2 (11)
Back, pain (Musculoskeletal and connective tissue disorders) | 3 (53)
Bone, pain (Musculoskeletal and connective tissue disorders) | 3 (54)
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Head/headache (General disorders) | 1 (1)
Joint, pain (Musculoskeletal and connective tissue disorders) | 3 (54)
Pain-other (General disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (54)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (54)
Renal/GU-other (Renal and urinary disorders) | 1 (14)

LIMITATIONS AND CAVEATS:
The study closed prematurely before the planned enrollment of 20 patients due to poor patient accrual. The patient population was highly selected, were likely to have had disease with an indolent natural history.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No